CLINICAL TRIAL: NCT03794466
Title: Quantification of Pain Relief With Gonadal Vein Embolization for Pelvic Congestion Syndrome
Brief Title: Quantify the Degree of Pain Relief of Pelvic Congestion Syndrome Following Gonadal Vein Embolization
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00143045
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Pelvic Congestive Syndrome; Pelvic Pain
Keywords: gonadal vein embolization
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective is to quantify the degree of pain relief in patients undergoing gonadal vein embolization with coils as well as identify clinical or imaging factors that are predictive of a positive response to treatment, or poor response to treatment.

DETAILED DESCRIPTION:
Chronic pelvic pain affects almost 40% of women during their lifetime. Pelvic congestion syndrome (PCS) accounts for up to 30% of those with chronic pelvic pain. The most common underlying cause of PCS is incompetence or obstruction of the gonadal veins, resulting in painful congestion of the pelvic and perineal venous vasculature. Medical treatment is first line, and aims to suppress ovarian function and induce vasoconstriction of the venous system. Unfortunately, efficacy and long-term pain relief from medical therapy is limited. Coil embolization of the gonadal veins has been shown to decrease pain in those affected by PCS, although the degree of relief has not yet been quantified.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Meet the clinical and imaging criteria for the diagnosis of PCS and have no contraindications to coil embolization of the gonadal veins.
* Patients who are treated with coil embolization of the gonadal veins in the Interventional Radiology division between October 1, 2018 to October 1, 2019.

Exclusion Criteria:

* Patients less than 18 years of age.
* Patients who are found to have an underlying cause of pelvic congestion syndrome unrelated to venous congestion and insufficiency. This includes, but is not limited to, nutcracker syndrome, or a mass resulting in extrinsic compression of the gonadal veins.
* Patients who have received prior surgical therapy for PCS, including bilateral salpingo-oophorectomy (TAH-BSO), gonadal vein resection, or gonadal vein ligation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Study Population: Women, 18 years of age and older, who are candidates for gonadal vein embolization in the Interventional Radiology division at the University of Kansas Medical Center from October 1, 2018 to October 1, 2019.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quantify pain relief using the Pelvic Congestion Symptom Pain Scale after gonadal vein embolization | Change from baseline (before gonadal vein embolization) to 360 days post-procedure.
  quantify the degree of pain relief in patients undergoing gonadal vein embolization with coils using a survey consisting 4 questions. Answers will be given values 0-4, which higher values are considered to be worse outcomes. One question is "On average, how many days a week do you experience pelvic pain?" Answers would be none (0), 1-2 days a week (1), 3-4 days a week (2), 5-6 days a week (3), and every day of the week (4). Maximum total amount of points will be 16. This is the number of points added together from all 4 questions.

SECONDARY OUTCOMES:
Predict positive or poor response to gonadal vein embolization treatment | Change from baseline (before gonadal vein embolization) to 360 days post-procedure.
  Identify clinical or imaging factors that are predictive of a positive response to treatment, or poor response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adam S Alli, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ignacio EA, Dua R, Sarin S, Harper AS, Yim D, Mathur V, Venbrux AC. Pelvic congestion syndrome: diagnosis and treatment. Semin Intervent Radiol. 2008 Dec;25(4):361-8. doi: 10.1055/s-0028-1102998. PMID 21326577
- [Background] O'Brien MT, Gillespie DL. Diagnosis and treatment of the pelvic congestion syndrome. J Vasc Surg Venous Lymphat Disord. 2015 Jan;3(1):96-106. doi: 10.1016/j.jvsv.2014.05.007. Epub 2014 Jun 25. PMID 26993690
- [Background] Koo S, Fan CM. Pelvic congestion syndrome and pelvic varicosities. Tech Vasc Interv Radiol. 2014 Jun;17(2):90-5. doi: 10.1053/j.tvir.2014.02.005. PMID 24840963
- [Background] Lopez AJ. Female Pelvic Vein Embolization: Indications, Techniques, and Outcomes. Cardiovasc Intervent Radiol. 2015 Aug;38(4):806-20. doi: 10.1007/s00270-015-1074-7. Epub 2015 Mar 25. PMID 25804635
- [Background] Daniels JP, Champaneria R, Shah L, Gupta JK, Birch J, Moss JG. Effectiveness of Embolization or Sclerotherapy of Pelvic Veins for Reducing Chronic Pelvic Pain: A Systematic Review. J Vasc Interv Radiol. 2016 Oct;27(10):1478-1486.e8. doi: 10.1016/j.jvir.2016.04.016. Epub 2016 Jul 7. PMID 27397619
- [Background] Brown CL, Rizer M, Alexander R, Sharpe EE 3rd, Rochon PJ. Pelvic Congestion Syndrome: Systematic Review of Treatment Success. Semin Intervent Radiol. 2018 Mar;35(1):35-40. doi: 10.1055/s-0038-1636519. Epub 2018 Apr 5. PMID 29628614
- [Background] Guirola JA, Sanchez-Ballestin M, Sierre S, Lahuerta C, Mayoral V, De Gregorio MA. A Randomized Trial of Endovascular Embolization Treatment in Pelvic Congestion Syndrome: Fibered Platinum Coils versus Vascular Plugs with 1-Year Clinical Outcomes. J Vasc Interv Radiol. 2018 Jan;29(1):45-53. doi: 10.1016/j.jvir.2017.09.011. Epub 2017 Nov 22. PMID 29174618

DOCUMENTS (1):
  • Study Protocol (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03794466/Prot_000.pdf